CLINICAL TRIAL: NCT04903236
Title: MR-BIO: a Study to Evaluate Changes in MR Imaging and Biological Parameters
Acronym: MR-BIO
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ananya Choudhury, Chair and Honorary Consultant in Clinical Oncology, University of Manchester
Other Study IDs: NHS001677
Record Dates: First submitted 2020-12-22; First posted 2021-05-26 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biospecimens collected and stored from each patient will include the following; tissue in the form of a diagnostic block in a Formalin Fixed Paraffin Embedded (FFPE) block, whole blood, plasma, and urine (both cell containing and cell depleted).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-patient healthy volunteer: Undertake MR Imaging to enable development of sequences.
- Patient: Provide weekly blood and urine samples during period of radiotherapy as well as additional MR images.

SUMMARY:
The MR BIO study aims to understand the changes in the tumour and normal tissues during a course of radiotherapy. This is accomplished by studying the MR images taken during each treatment session on the MR Linear accelerator (MR Linac). The overarching hypothesis is that changes in MR imaging and biological parameters from blood, tissue, or urine biomarkers can be measured during radiotherapy and associated with clinical outcome.

The MR Linac is a new radiotherapy machine with an on board MR scanner. This enables us to take images with high resolution and target the tumours more precisely and also reduce the dose to normal tissues. All patients undergoing treatment in the MR Linac at the Christie hospital will be considered for enrolment regardless of tumour site being treated.

The study participants will receive the standard of care treatment for their disease condition. In addition, they will be requested to give weekly blood and urine samples during the course of radiotherapy and at first follow up. On completion of radiotherapy treatment, the participants will continue to be on standard of care follow up protocol with the treating oncologist.

A small cohort of ten healthy volunteers will also be recruited to the study to develop and select some of the MR sequences only; they will not provide blood or urine samples. The healthy volunteers will be scanned for no more than one hour per session for a maximum of two sessions in total. These optimised sequences can then be used in the patient cohort.

ELIGIBILITY:
Inclusion Criteria:

Be willing and able to provide written consent. Over 18 years of age. Undergo and satisfy MRI Safety Screening Patient volunteers must be under the care of a clinical oncologist at The Christie NHS Foundation Trust and be planned to receive radiotherapy to the target site to be imaged.

Patient volunteers must be able to give blood and/or urine sample as required through the treatment period.

Non-patient (healthy) volunteers must have no known or suspected significant medical condition.

Exclusion Criteria:

The following apply to both patients and healthy volunteers:

Any conditions that would be a contra-indication to MRI including:

* Failure to satisfy MRI Safety Screening Form
* Implanted pacemakers and/or pacing wires
* Cochlear implants
* Programmable hydrocephalus shunts
* Ferromagnetic implants
* Unable to tolerate MR scans
* Known HIV or active HepB or C
* Pregnancy Healthy volunteers must not be a member of the study team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Christie.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of biomarkers | Up to five years
  Analysis of MR images will be performed using in-house protocols based on established mathematical modelling techniques. Pearson correlation analysis will be used to assess relationships between MRI parameters and tissue markers. For oxygen enhanced imaging, two-sample unpaired t-tests will be used to identify changes in tissue oxygen in MR images. Descriptive statistics will be presented using median and 95% confidence intervals (CI) or standard deviation (SD). In addition, Bland-Altman analysis will be performed to calculate bias and 95% limits of agreement between the two measurement techniques.

SECONDARY OUTCOMES:
Correlation with patient reported toxicity | Up to five years
  Association of detected imaging changes with variations in patient-reported toxicity and radiotherapy response at first follow up after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ananya Choudhury, PhD, FRCR, MRCP, MA, MB BChir,, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No